CLINICAL TRIAL: NCT01138891
Title: Sonication of Explanted Breast Implants for Detection of Subclinical Infection
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: University Hospital, Basel, Switzerland (Other); Medical University Innsbruck (Other); Clinic Löwencenter, Luzern, Switzerland (Unknown); Clinic Birshof, Münchenstein, Switzerland (Unknown); Crossklinik im Merian Iselin Spital, Basel, Switzerland (Unknown)
Responsible Party: Dr. Andrej Trampuz, University Hospital Lausanne, Switzerland
Other Study IDs: EKBB_2008
Record Dates: First submitted 2010-06-07; First posted 2010-06-08 (Estimated); Last update posted 2010-06-09 (Estimated); Status verified 2010-06

CONDITIONS: Implants, Breast
Keywords: Breast implants; capsular contraction; sonication; biofilm; Complications; surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Breast implants
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Removed breast implants for any reason

SUMMARY:
Objective. Capsular contracture is a frequent complication after breast implantation with unclear etiology.

Summary Background Data: Microorganisms may trigger chronic periimplant inflammation with subsequent capsular fibrosis.

Study Hypothesis: The investigators hypothesize that with sonication adherent microorganisms can be detected on removed implants .

Methods: In a prospective multicentre study all breast implants explanted are collected to be analyzed by sonication. The resulting culture results are correlated with patient, surgical and implant characteristics.

DETAILED DESCRIPTION:
The study is performed in order to find a correlation between the degree of capsular fibrosis and presence of biofilm bacteria on the surface of the implant.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or more
* Undergoing breast implant removal for any reason at one of the participating center
* Explantation of breast implant performed between February 2006 and March 2009

Exclusion Criteria:

* Obvious contamination of the breast implant in the operating room or during transportation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Five plastic surgery clinics in Switzerland participated in this study (Basel, Luzern, Dornach, Lausanne, Münchenstein).
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2006-02; Primary Completion 2009-03 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich M Rieger, MD, Principal Investigator — Department of Plastic, Reconstructive & Aesthetic Surgery, Medical University, Innsbruck, Austria

REFERENCES:
- [Background] Rieger UM, Pierer G, Luscher NJ, Trampuz A. Sonication of removed breast implants for improved detection of subclinical infection. Aesthetic Plast Surg. 2009 May;33(3):404-8. doi: 10.1007/s00266-009-9333-0. Epub 2009 Mar 26. PMID 19322605
- [Derived] Rieger UM, Mesina J, Kalbermatten DF, Haug M, Frey HP, Pico R, Frei R, Pierer G, Luscher NJ, Trampuz A. Bacterial biofilms and capsular contracture in patients with breast implants. Br J Surg. 2013 May;100(6):768-74. doi: 10.1002/bjs.9084. Epub 2013 Mar 6. PMID 23468161